CLINICAL TRIAL: NCT07207356
Title: The Efficacy of Ultrasound Guided Transcutaneous Pulsed Radiofrequency for Cervical Radiculopathy: a Randomized, Sham-controlled, Double-blind Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20250724R
Record Dates: First submitted 2025-10-01; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Cervical Radiculopathy
Keywords: cervical radiculopathy; pulsed radiofrequency; transcutaneous pulsed radiofrequency; ultrasound guided
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- true transcutaneous pulsed radiofrequency group (Experimental)
  Interventions: Device: true transcutaneous pulsed radiofrequency
- Sham transcutaneous pulsed radiofrequency group (Sham Comparator)
  Interventions: Device: Sham device

INTERVENTIONS:
Device: true transcutaneous pulsed radiofrequency — participants will receive ultrasound guidance to localize the target cervical nerve root (e.g., C5-C7) before treatment. A high-frequency linear transducer will be used with the patient in a sitting position. Transcutaneous pulsed radiofrequency (TCPRF) will be applied using the StimOn™ Pain Relief System (GM2439, Gimer Medical Co., Ltd, Taiwan; FDA 510(k) No. K213802). The device delivers a 500-kHz symmetric biphasic sine wave at 2 Hz with a 25-ms pulse. Each session lasts 30 minutes, divided into two 15-minute phases, with treatment administered 3 times per week for 4 weeks (12 sessions in total).
  Arms: true transcutaneous pulsed radiofrequency group
Device: Sham device — participants will receive ultrasound guidance to localize the target cervical nerve root (e.g., C5-C7) before treatment. A high-frequency linear transducer will be used with the patient in a sitting position. Sham device will be applied. No active current will be delivered. Each session lasts 30 minutes, divided into two 15-minute phases, with treatment administered 3 times per week for 4 weeks (12 sessions in total).
  Arms: Sham transcutaneous pulsed radiofrequency group

SUMMARY:
Cervical radiculopathy (CR) is a painful condition caused by irritation of the cervical nerve roots, often leading to neck, shoulder, and arm pain, sometimes with numbness or weakness. These symptoms can reduce quality of life and place a burden on healthcare systems. Current treatments, such as physical therapy, cervical traction, and medication, are often not fully effective. Pulsed radiofrequency (PRF) has shown benefits for nerve-related pain, but because it requires an invasive procedure, its use is limited.

Transcutaneous pulsed radiofrequency (TCPRF) is a non-invasive version of PRF. It has shown promising results in animal studies and in clinical research for knee and shoulder conditions, but has not been tested for CR. Recent improvements in ultrasound allow more precise targeting of cervical nerve roots, making ultrasound-guided TCPRF a potentially safe and accessible treatment option.

This pilot study will evaluate the efficacy and safety of ultrasound-guided TCPRF in patients with CR compared to a sham treatment. A total of 32 participants with CR lasting more than six weeks will be randomly assigned to either TCPRF or sham treatment. Both groups will receive 12 treatment sessions over four weeks, combined with a standard rehabilitation program.

The main outcome is pain intensity measured by the Numeric Rating Scale (NRS). Secondary outcomes include neck-related disability, medication use, and any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 75 years old.
* Clinical diagnosis of cervical radiculopathy, defined by:

  1. Presence of neck pain or paresthesia radiating to the unilateral upper extremity with radicular and dermatomal pattern;
  2. Positive Spurling's test;
  3. Positive cervical distraction test
* Symptoms lasting for over 6 weeks
* Numeric Rating Scale (NRS) for arm pain ≥ 4 out of 10
* MRI or CT-confirmed nerve root compression, corresponding to clinical symptoms.
* Able to provide written informed consent and comply with study procedures

Exclusion Criteria:

* History of cervical spine surgery.
* Motor deficit on involving limb
* Presence of axial neck pain without radicular symptoms
* Symptoms from shoulder, elbow, or wrist joint or other musculoskeletal co-morbidity such as rheumatologic disease or carpal tunnel syndrome
* Evidence of serious underlying pathology (e.g., tumor, infection, fracture, or myelopathy)
* Prior exposure to epidural steroid injection or pulsed radiofrequency therapy within the past 6 months
* Presence of pregnancy or breastfeeding.
* History of epilepsy or electronic devices implanted in the body
* Active infection or skin disease at the stimulator contact site
* Allergy to electrode patch
* Unable to understand the study protocol or provide written

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | baseline, at the end of week 2, at the end of week 4 (post-treatment), and at a 3-month follow-up after the intervention
  Participants will rate their average pain over the past week on a scale from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | baseline, at the end of week 2, at the end of week 4 (post-treatment), and at a 3-month follow-up after the intervention
  The NDI consists of ten items. These include seven questions related to daily functional activities, two addressing symptom severity, and one focused on concentration. The total score is calculated by summing the responses to all items, with higher scores reflecting greater levels of disability. According to Vernon et al, scores of 0-4 indicate no disability, 5-14 indicate mild disability, 15-24 moderate disability, 25-34 severe disability, and scores above 35 reflect complete disability.
medication usage | baseline, at the end of week 2, at the end of week 4 (post-treatment), and at a 3-month follow-up after the intervention
  During the intervention and follow-up period, participants who experience unbearable pain will be allowed to take rescue medication, consisting of 500 mg of oral acetaminophen up to four times per day. The frequency and amount of rescue medication used will be documented at each assessment point.

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided